CLINICAL TRIAL: NCT02718651
Title: Identification of Response to ALK-targeted Treatment in Lung Cancer Patients by Monitoring Tumor DNA in Blood Samples
Brief Title: Blood-based Identification and Monitoring of Patients With ALK-translocated Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1881-2; 1-10-72-266-15 (Other: The National Committee on Health Research Ethics); 1-16-02-56-16 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2016-03-18; First posted 2016-03-24 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2016-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: ALK rearrangement; Circulating tumor DNA; Plasma DNA; Non-small cell lung cancer; Tyrosine kinase inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples - plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Genetic rearrangements in the Anaplastic Lymphoma Kinase (ALK) gene result in the creation of a variety of oncogenic fusion proteins that drive malignancy in a subset of non-small cell lung cancers (NSCLC) patients. Treatment with the ALK small tyrosine kinase inhibitor (TKI) crizotinib has produced remarkable results for ALK-positive patients, however the current diagnostic tests used in the clinic are not sufficiently detailed and require a tumor biopsy.

The aim of this study is to use a new diagnostic test to detect ALK rearrangements using next generation sequencing, which will improve the diagnosis and treatment of ALK-positive NSCLC patients. Furthermore, this test will be performed on blood samples, making it minimally invasive for the patients. It is our believe that circulating tumor DNA (ctDNA) in blood can be employed as an easy accessible and comprehensive source of information to diagnose ALK-positive disease, but also as a means of monitoring patient response during treatment. Quantitation of the the amount of ALK rearrangement will give information about which patients benefit from treatment and when treatment is no longer effective. The project will be a multicenter study where blood samples will be collected every 6 weeks from patients treated at four major hospitals in Denmark.

This study will benefit future patients with lung cancer, as it will improve both the monitoring and evaluation of their treatment. Monitoring patients during treatment will provide more knowledge of disease progression and the effect of ALK-TKI treatment, contributing to a greater selection of patients, who will respond to treatment. This will potentially allow effective treatment to continue longer than with conventional methods

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer diagnosis
* Biopsy-verified ALK-translocation

Exclusion Criteria:

* Patients were it is not possible to retrieve a biopsy
* Patients with squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALK-translocated lung cancer
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Meldgaard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No